CLINICAL TRIAL: NCT01325116
Title: Delayed Educational Reminders for Long-term Medication Adherence in ST-Elevation Myocardial Infarction (DERLA-STEMI): Cluster-randomized Controlled Trial
Brief Title: Delayed Educational Reminders in Acute Myocardial Infarction (MI)
Acronym: DERLA-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jon-David Schwalm, Interventional Cardiologist, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MAC-DS-03-2011
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Acute Myocardial Infarction; STEMI
Keywords: STEMI; Medication Adherence; Quality Improvement
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Usual post-STEMI care
  Interventions: Behavioral: Educational Reminder
- Intervention (Experimental): Recurrent, personalized, educational reminders sent via post on behalf of the interventional cardiologist to the patient and their family physician urging long-term adherence to secondary prevention medications post-STEMI. A copy of the letter will be provided to the patient to take to their pharmacist.
  Interventions: Behavioral: Educational Reminder

INTERVENTIONS:
Behavioral: Educational Reminder — Personalized letters sent via post to the patient and their family physician at one, five, eight, and eleven months after their angiogram, sent on behalf of the interventional cardiologist. The patient letter provides a review of the role of each of the cardiac medications and urges long-term adherence. The language in the patient letter is simplified to a grade 6 level; this letter was tested for understanding and acceptability amongst a series of Cardiology patients.At the same time, close examination of data from Ontario indicated large stepwise declines in adherence at 30 and 60 days post-STEMI. To address this, patients will be provided an additional postcard type reminder two months post-STEMI.

SUMMARY:
ST segment elevation myocardial infarction (STEMI) is a common presentation of heart attack constituting approximately 30% of all cases. Clinical guidelines around the world support the prolonged use of secondary preventative medications including aspirin, clopidogrel, statin, beta-blocker and angiotensin blockers with the highest recommendations. While in-hospital and discharge prescription rates are excellent, adherence to these essential life-saving medications is far less than ideal, even a few months following hospital discharge. The investigators plan to capitalize on the existing structure of the SMART-AMI project already underway in LHIN IV to undertake a randomized controlled trial evaluating a reminder sent on behalf of the interventional cardiologists, delivered by mail, at 1, 2, 5, 8, and 11-months post-discharge, reviewing the evidence for life-saving cardiac medications and urging long-term adherence to secondary preventative cardiac medications. This will be sent to the family physician and the patient, using audience-appropriate language. If the DERLA-STEMI project is accepted by physicians and patients, found to be both feasible and effective, then this simple and low-cost intervention will be studied in all patients with an abnormal coronary angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with STEMI to a hospital in LHIN IV, coronary angiogram with and without PCI at Hamilton General Hospital during hospital admission

Exclusion Criteria:

* Non-english speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cardiac Medication Use | 3 and 12 months
  Proportion of patients who report taking all cardiac medication classes, measured three and twelve months post-STEMI. Specifically, we will assess whether patients are taking a statin, beta-blocker, angiotensin modifier (ACE or ARB), and aspirin at twelve months, and whether they are taking these plus a secondary antiplatelet (clopidogrel, prasugrel, or ticagrelor) at three months.

SECONDARY OUTCOMES:
Other Evidence-based Cardiac Medication Use | 3 and 12 months
  Proportion of patients who report actively taking aspirin, clopidogrel, statin, beta-blocker, and/or angiotensin blocker
Statin Dose | 3 and 12 months
  Proportion of patients taking high dose statins at three and twelve months
Medication Side-effects | 3 and 12 months
  Proportion of patients who report stopping medications due to side effects at three and twelve months
Discussion with Family physician/specialist | 3 and 12 months
  Proportion of patients who state that they had a discussion with their FP regarding the benefits of certain medications to prevent future heart attacks or that focused on medication compliance since their heart attack.
Use of medication combinations | 3 and 12 months
  The proportion of patients using 1 of 5, 2 of 5, 3 of 5, 4 of 5, or 5 of 5 medications at three and twelve months.
Adherence | 3 and 12 Months
  Proportion of patients with a perfect Morisky Green Levine Test for cardiac medication compliance at three and twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David R Schwalm, BSc, MD, Principal Investigator — McMaster University/Hamilton Health Sciences/Population Health Research Institute
Locations (1):
- Hamilton Health Sciences-General Site, Heart Investigation Unit, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Schwalm JD, Ivers NM, Natarajan MK, Taljaard M, Rao-Melacini P, Witteman HO, Zwarenstein M, Grimshaw JM. Cluster randomized controlled trial of Delayed Educational Reminders for Long-term Medication Adherence in ST-Elevation Myocardial Infarction (DERLA-STEMI). Am Heart J. 2015 Nov;170(5):903-13. doi: 10.1016/j.ahj.2015.08.014. Epub 2015 Aug 20. PMID 26542498
- [Derived] Ivers NM, Schwalm JD, Grimshaw JM, Witteman H, Taljaard M, Zwarenstein M, Natarajan MK. Delayed educational reminders for long-term medication adherence in ST-elevation myocardial infarction (DERLA-STEMI): protocol for a pragmatic, cluster-randomized controlled trial. Implement Sci. 2012 Jun 9;7:54. doi: 10.1186/1748-5908-7-54. PMID 22682691